CLINICAL TRIAL: NCT05476874
Title: Clinical Study on Improvement of Peritoneal Catheter Placement in Ventriculoperitoneal Shunt Surgery With a Splitable Trocar
Brief Title: Improvement of Peritoneal Catheter Placement in VPS With a Splitable Trocar
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Zhen-Zhou Chen, Clinical Professor, Southern Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJH-003
Record Dates: First submitted 2022-07-21; First posted 2022-07-27 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Hydrocephalus
Keywords: Hydrocephalus; Ventriculoperitoneal Shunt; Distal shunt failure; Trocar; Complications
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Mini-laparotomy Group (OLG) (Active Comparator): Distal shunt placement through open mini-laparotomy.
  Interventions: Procedure: Open Mini-Laparotomy
- Abdominal Puncture Group （APG） (Experimental): Distal shunt placement through abdominal puncture.
  Interventions: Procedure: Abdominal Puncture

INTERVENTIONS:
Procedure: Open Mini-Laparotomy — A 5-cm paraumbilical skin is made, and the abdominal wall is incised in layers. The distal catheter tip is inserted into the peritoneal cavity in a craniocaudal direction, and the abdominal wound is sutured in layers.
  Arms: Open Mini-laparotomy Group (OLG)
Procedure: Abdominal Puncture — An about 0.5-cm paraumbilical incision made to allow introduction of a splitable trocar. The trocar is pierced through the abdominal wall into the abdominal cavity. Pull out the puncture cone, and adjust the trocar towards the pelvis. The distal catheter tip is inserted into the peritoneal cavity through the puncture cannula. Then the splitable puncture cannula is split apart and removed. The skin incision requires only one stitch.
  Arms: Abdominal Puncture Group （APG）

SUMMARY:
This study is a phase I/IIa, single-center, open-labeled, randomized, controlled clinical trial. The aim of this study is to evaluate the safety and efficacy of a modified ventriculoperitoneal catheter placement using a splitable trocar for ventriculoperitoneal shunt.

DETAILED DESCRIPTION:
This study is a phase I/IIa, single-center, open-labeled, randomized, controlled clinical trial. Patients hospitalized with hydrocephalus will be enrolled and randomly allocated into open mini-laparotomy group (OLG) or abdominal puncture group (APG) for insertion of the peritoneal catheter. Observe will followed for up to at least 6 months after surgery. The primary endpoint is the rate of overall shunt complication or failure within the first 6 months after surgery, and duration of the abdominal catheterization. The secondary endpoints are rate of distal shunt failure, the overall incidence of various adverse reactions, abdominal incision size, analgesic use as evaluated on Day 5 postoperatively, duration of hospital stay. Moreover, neurological function of patients (mRS, maxillary hydrocephalus scale) and CT measurement of Even index will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older with new-onset hydrocephalus, including obstructive hydrocephalus, traffic hydrocephalus and special types of hydrocephalus, normal pressure hydrocephalus (NPH), idiopathic intracranial hypertension (IIH), benign intracranial hypertension, pseudotumor cerebri, etc., regardless of gender.
2. Initial diagnosis of hydrocephalus requiring ventriculoperitoneal shunt or shunt failure requiring secondary surgery to replace the shunt.
3. Provided written informed consent.

Exclusion Criteria:

1. Previous abdominal surgery (except ventriculoperitoneal shunt).
2. Pregnancy
3. Peritonitis
4. Patients with cognitive impairment and inability to communicate.
5. Expected survival less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of shunt failure | 6 months
  Overall rate of shunt failure requiring revision
Duration of the abdominal catheterization | During the surgery
  Duration of the abdominal catheterization, defined as the time from abdominal incision to abdominal skin suture completed.

SECONDARY OUTCOMES:
Rate of distal shunt failure | 6 months
  Rate of distal shunt failure requiring revision
The incidence of adverse reactions | 6 months
  The overall incidence of various adverse reactions
Abdominal incision size | During the surgery
  Abdominal incision size
The incidence of anargesic drug use | Day 5 after surgery
  The incidence of anargesic drug use as evaluated on day 5 postoperatively
Duration of hospita stay | During perioperative period
  Duration of hospita stay, defined as day of admission until discharge from the neurosurgical ward.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen-Zhou Chen, Dr., Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schucht P, Banz V, Trochsler M, Iff S, Krahenbuhl AK, Reinert M, Beck J, Raabe A, Candinas D, Kuhlen D, Mariani L. Laparoscopically assisted ventriculoperitoneal shunt placement: a prospective randomized controlled trial. J Neurosurg. 2015 May;122(5):1058-67. doi: 10.3171/2014.9.JNS132791. Epub 2014 Dec 23. PMID 25534231
- [Result] Gravbrot N, Aguilar-Salinas P, Walter CM, Dumont TM. Laparoscopically Assisted Ventriculoperitoneal Shunt Placement Is not Cost-Effective nor Preventive for Distal Shunt Malfunction. World Neurosurg. 2020 May;137:e308-e314. doi: 10.1016/j.wneu.2020.01.193. Epub 2020 Feb 3. PMID 32028009
- [Result] Lou M, Zhou G, Zhao Y. The application of improved abdominal wall punctures technique in ventriculoperitoneal shunt for hydrocephalus: a retrospective analysis versus open mini-laparotomy. Br J Neurosurg. 2018 Dec;32(6):650-652. doi: 10.1080/02688697.2018.1429564. Epub 2018 Jan 24. PMID 29363332